CLINICAL TRIAL: NCT02764879
Title: Effect of Omega 3 Fatty Acids on Chronic Periodontitis Patients in Postmenopausal Women: A Randomized Controlled Clinical Study
Brief Title: Effect of Omega 3 on Periodontitis in Postmenopausal Women
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: October 6 University (Other)
Responsible Party: Principal Investigator, Enas Elgendy, Ass. Prof., October 6 University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 3
Record Dates: First submitted 2016-05-03; First posted 2016-05-06 (Estimated); Last update posted 2016-05-06 (Estimated); Status verified 2016-05

CONDITIONS: Chronic Periodontitis
Keywords: Omega 3 fatty acids; Root planning; chronic periodontitis
MeSH Terms: conditions — Chronic Periodontitis | interventions — Fatty Acids, Omega-3; Docosahexaenoic Acids; Tooth Exfoliation; Root Planing

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- omega 3 group (Experimental): scaling and root planing omega3 received 2 times daily-for 6 months
  Interventions: Dietary Supplement: Omega 3 fatty acids; Procedure: scaling and root planing
- control group (Placebo Comparator): scaling and root planing placebo soft gelatin capsules 2 times daily-for 6 months
  Interventions: Procedure: scaling and root planing; Other: placebo soft gelatin capsules

INTERVENTIONS:
Dietary Supplement: Omega 3 fatty acids — omega3 received 2 times daily-for 6 months
  Other Names: omega 3
  Arms: omega 3 group
Procedure: scaling and root planing
Other: placebo soft gelatin capsules — placebo soft gelatin capsules received 2 times daily-for 6 months
  Arms: control group

SUMMARY:
The study was aimed to investigating changes in periodontal parameters and superoxide dismutase activity after root surface debridement with and without Omega 3 fatty acids (ω-3 FAs) supplementation in postmenopausal women. Adjunctive Omega 3 fatty acids supplements reduce periodontal inflammation and improve the status of systemic enzymatic antioxidants in postmenopausal women.

DETAILED DESCRIPTION:
Fifty postmenopausal women with chronic periodontitis were divided randomly into two groups: Group 1 (n=25) were provided periodontal treatment in the form of scaling and root planing (SRP) plus placebo soft gelatin capsules while group 2 (n=25): patients were received SRP along with systemic administration of Omega 3 fatty acids. Clinical parameters and superoxide dismutase (SOD) activity in the gingival crevicular fluid were recorded at baseline, 3 and 6 months after therapy. The research has been conducted between July 2014 and June 2015. By the end of the study period, the Omega 3 treated group was able to achieve a greater mean probing pocket depth reduction, mean gain in clinical attachment level, as well as greater increase in SOD activity (P<0.01) compared to SRP alone.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women with generalized chronic periodontitis (clinical attachment loss more than 30% of the teeth)
* With probing pocket depth ≥ 5mm.
* The age ranged between 45 and 60 years (To avoid the wide variation between individual cases in order to make the sample more homogeneous. Furthermore elderly patients above 60 years are usually not willing to have periodontal treatment).
* Postmenopausal status for at least 1 year.
* Presence of at least six teeth in the mouth.

Exclusion Criteria:

* Any systemic disease that affect the periodontium.
* Women who take anti-inflammatory drugs, antibiotics or vitamins within the previous 3 month.
* Women who use mouth washes regularly
* Smoking
* History of alcohol abuse
* Participation in other clinical trials.
* Obese women (Body mass index (BMI) ≥ 30).

Ages: 45 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2014-07; Primary Completion 2015-01 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
superoxide dismutase (SOD) activity in the gingival crevicular fluid | up to 6 months
  Superoxide dismutase activity in the gingival crevicular fluid was carried out at baseline, 3 and 6 months post treatment.

SECONDARY OUTCOMES:
Plaque Index | up to 6 months
  plaque index was recorded at baseline and at 3 and 6 months post treatment.
Gingival index | up to 6 months
  Gingival index was recorded at baseline, 3, 6 months post treatment
Probing pocket depth | up to 6 months
  Probing pocket depth in mm was recorded at baseline, 3, 6 months treatment
Clinical attachment level | up to 6 months
  Clinical attachment level was recorded at baseline, 3 and 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Enas A Elgendy, MD, Principal Investigator — October University

IPD SHARING:
Plan to Share IPD: No